CLINICAL TRIAL: NCT02466048
Title: Clinical Trial to Evaluate the Efficacy and Safety of SurgiFill™ on Spinal Fusion -Comparison Between Autograft Mixed With SurgiFill™ and Autograft in Spinal Fusion-
Brief Title: Efficacy and Safety of SurgiFill™ on Spinal Fusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sewon Cellontech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02SGF
Record Dates: First submitted 2015-06-01; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Spinal Fusion Acquired; Fusion of Spine (Disease)
Keywords: spinal fusion; bone graft; collagen
MeSH Terms: conditions — Disease | interventions — Spinal Fusion; Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SurgiFill™ on Spinal Fusion (Experimental): In one side of one patient, autogenous bones and SurgiFill™ will be grafted; and in the other side, only the autogenous bones will be grafted.
  Interventions: Procedure: Spinal Fusion; Device: SurgiFill™
- Autograft on Spinal Fusion (Active Comparator): In one side of one patient, autogenous bones and SurgiFill™ will be grafted; and in the other side, only the autogenous bones will be grafted.
  Interventions: Procedure: Spinal Fusion

INTERVENTIONS:
Procedure: Spinal Fusion — Spinal fusion, also known as spondylodesis or spondylosyndesis, is a surgical technique used to join two or more vertebrae. Supplementary bone tissue, from the patient (autograft), is used in conjunction with the body's natural bone growth (osteoblastic) processes to fuse the vertebrae. Either the right or left side of one patient will be selected for the study group, and the other, for the control group, through randomization. In the study group site, SurgiFill™ and the autogenous bone mixture shall be transplanted, whereas in the control group site, only the autogenous bone shall be transplanted. The autogenous bones are from iliac part.
  Other Names: Spinal Fusion, spondylodesis, spondylosyndesis, bone graft
Device: SurgiFill™ — SurgiFill™ is a gel-type high-purity ateolcollagen for bone grafting. SurgiFill™ is used with autogenous iliac graft for dorsolateral spinal fusion.
  Arms: SurgiFill™ on Spinal Fusion

SUMMARY:
This study was designed to investigate the safety and efficacy of SurgiFill™, a bone grafting material, in patients with spinal fusion.

DETAILED DESCRIPTION:
This study is an open-trial study. The study will be explained to the subjects and they voluntarily agreed to participate in it. Their eligibility to participate in the study will be checked, either the right or left side of one patient will be selected for the study group, and the other, for the control group, through randomization. In the area for the study group, autogenous bones and SurgiFillTM will be grafted; and in the area for the control group, only the autogenous bones will be grafted. They will be asked to follow the guidelines of the investigators during the study and to visit the hospital seven times, including for screening. At each visit, the subjects undergo an examination with doctors, a CT scan, a X-ray, and a SPECT/CT procedure to evaluate the safety and efficacy of SurgiFill™. (*If the subject gets surgery on the screening date, the total number of his or her visits will be six).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who require spinal fusion
2. Adult patients aged 20 or older
3. Patients who voluntarily agreed to participate in this study and signed the informed consent form, and who do not fall into any of the exclusion criteria

Exclusion Criteria:

1. Patients or their family members with a history of an, or an ongoing, autoimmune disease
2. Patients with a history of anaphylactic response
3. Patients with hypersensitivity to grafting materials
4. Patients with hypersensitivity to pig protein
5. Patients with osteomyelitis in the surgery area
6. Patients who are pregnant, breastfeeding, or planning to become pregnant
7. Patients with other tumors or a non-curable disease
8. Patients with a history of radiation therapy or cancer treatment within two years (Those who show normal or insignificant test results may be enrolled in this study and receive the SurgiFill™ injection based on the investigator's judgment.)
9. Patients with diabetes (Those who maintain a normal blood sugar level and did not develop complications may receive the SurgiFill™ injection based on the investigator's judgment, but the doctor's confirmation is required.)
10. Patients with an infection that required hospitalization for antibiotics or the administration of antiseptic agents
11. Patients who have been undergoing adrenocortical hormone therapy (Those who show normal or insignificant test results may be enrolled in this study and receive the SurgiFill™ injection based on the investigator's judgment.)
12. Patients with liver, heart, or kidney disease (Those who show normal or insignificant test results may be enrolled in this study and receive the SurgiFill™ injection based on the investigator's judgment. Hypertension patients are allowed.)
13. Patients who had been infected with a virus (Those who show normal or insignificant test results may be enrolled in this study and receive the SurgiFill™ injection based on the investigator's judgment.)
14. Patients with chronic renal failure or an endocrine system disease (Those who show normal or insignificant test results may be enrolled in this study and receive the SurgiFill™ injection based on the investigator's judgment.)
15. Patients who are considered inappropriate for participation in this study due to their condition (e.g., a mental illness) based on the investigator's judgment
16. Patients who had participated in another clinical trial (limited to those who participated in other studies on fracture within the last six months.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-10 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Volume change of bony fusion mass in the CT | 1week, 6month, and 12month
  A CT scan shall be conducted one week, and six and 12 months, post-operatively to calculate and record the bone integration volume. The changes in the bone integration volume shown in the CT images shall be compared and analyzed. In other words, the mean values of the experiment group's bone integration volume shown in CT images 1week, six and 12 months post-operatively shall be compared and analyzed.

SECONDARY OUTCOMES:
Degree change of bony fusion mass in the X-ray | 1month, 3month, 6month, and 12month
  A radiography shall be conducted one, three, six, and 12 months post-operatively, and at the additional unscheduled visits, and the PIs from different institutions (i.e., the Seoul St. Mary's PI and the Daejon St. Mary's PI) shall cross-evaluate the results. The mean values of the experiment group's surgical site bone integration level shown in X-ray images one, three, six and 12 months post-operatively shall be compared and analyzed.
Value of ROI(Region of interest) in the SPECT/CT | 3month
  The osteoblastic activity levels at the surgical sites of the experiment and control groups shall be compared at three months post-operatively.
VAS Score change of Back pain questionnaire | screening, 6month and 12 month
  The level of the pain (i.e., the lumbar pain and the pain radiating to the upper and lower extremities) shall be recorded using the VAS before the spondylodesis, and at six and 12 months post-operatively.
ODI Score change of Back pain questionnaire | screening, 6month and 12 month
  Using the ODI score from the ODQ, the disturbances in the daily activities associated with the lumbar pain shall be compared before the spondylodesis, and at six and 12 months post-operatively.

OTHER OUTCOMES:
Number of abnormal blood test result of participants with adverse events as a measure of safety | up to 12month
  Regardless of the clinical trial, if there are blood tests' results of participants with adverse events such as hematologic examination (WBC, RBC, Hemoglobin(Hb), Hematocrit(Hct), Platelet(PLT), ESR) and general chemistry (BUN, Creatinine(Cr), AST, ALT, CRP) closed to the day of regular visit, they shall be recorded on the CRF at screening or after spinal fusion. If there is any abnormality of the results, the number of abnormal blood test result will be recorded, and then additionally the result shall be analyzed according to the investigator's judgment.

CONTACTS AND LOCATIONS:
Overall Officials: Young Hoon Kim, MD, Principal Investigator — The Catholic Univ. of Korea, Seoul St. Mary's Hospital; Young Yul Kim, MD, Principal Investigator — The Catholic Univ. of Korea, Daejeon St. Mary's Hospital
Locations (2):
- South Korea (2):
  - The Catholic Univ. of Korea, Daejeon St. Mary's Hospital, Daejeon, Daejeon
  - The Catholic Univ. of Korea, Seoul St. Mary's Hospital, Seoul, Seoul